CLINICAL TRIAL: NCT03713645
Title: Dosing Strategies for de Novo Once-daily Extended Release Tacrolimus (LCPT) in Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 25286
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Results first posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-04

CONDITIONS: Kidney Transplant
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tacrolimus extended-release 0.13mg/kg/day (Experimental): Tacrolimus extended-release is initiated within post-operative day 3 of kidney transplant
  Interventions: Drug: Tacrolimus Extended Release Oral Tablet [Envarsus] 0.13mg/kg/day initiated within post-operative day 3 after kidney transplant

INTERVENTIONS:
Drug: Tacrolimus Extended Release Oral Tablet [Envarsus] 0.13mg/kg/day initiated within post-operative day 3 after kidney transplant — Study drug (tacrolimus extended-release) initiated at 0.13/mg/kg/day for all patients

SUMMARY:
Outcomes after kidney transplantation have been significantly enhanced with the advances made in immunosuppressive therapies. Tacrolimus is currently marketed as an extended-release once-daily formulation dosing option for patients, decreasing pill burden and possibly decreasing adverse effects. Some transplant recipients have been shown to have higher dosage requirements. According to the literature, this can be linked to genetic disparities in the metabolism of tacrolimus.. This potential complication, where differences on specific genes alters metabolism of tacrolimus, can increase difficulty in getting to a therapeutic drug level for immunosuppresants and is one large factor that contributes to the fact that kidney transplant survival rates differ between patients. Due to the enhanced bioavailability of Meltdose formulation once-daily extended-release tacrolimus, its de novo use in recent research and practice has been shown to expedite achievement of target tacrolimus trough concentrations. De novo use of once-daily tacrolimus formulations is understudied. Through a prospective investigational study, we aim to determine the optimal strategy for de novo dosing of once-daily extended release tacrolimus (MeltDose formulation) for kidney transplant recipients at Temple University Hospital.

DETAILED DESCRIPTION:
Patients will be identified when an organ from live or deceased donor becomes available for kidney transplant. Prior to receiving their kidney transplant, subjects will be screened for inclusion/exclusion criteria on the day of transplantation. During the pre-operative preparation for transplant, patients will be consented for surgery and consented for the study at the same time if they volunteer to be included. The transplant surgeon performing the transplant operation will be responsible for screening the patients for inclusion and exclusion criteria as well as obtaining informed consent. Patients will need to provide informed consent to be included in the study, and will receive a copy of their consent. Each potential participant will be approached by the transplant surgeon and informed of all information pertinent to the study prior to providing consent. No advertisements for recruitment will be performed and no compensation will be provided for participation.

This study is a single center prospective observational study conducted at Temple University Hospital (TUH). All participants will be consented for all procedures involved in this study. This study will utilize the QUEST questionnaire (attached) to evaluate the severity of tremors at 1 month. Data to be collected includes tacrolimus trough levels, study drug dosing, hemoglobin A1c, incidence and severity of tremors, potassium, glomerular filtration rate, and rejection episodes.

Day 0 Study drug (tacrolimus) initiated at 0.13/mg/kg/day for all patients (the day of initiation decided per transplant surgeon discretion)

Day 0-4 Inpatient laboratory parameters checked every 24 hours (serum creatinine, tacrolimus level, glomerular filtration rate, potassium, blood glucose)

Day 4-30 Outpatient laboratory parameters checked three times weekly on Monday, Wednesday, and Friday (serum creatinine, tacrolimus level, glomerular filtration rate, potassium, blood glucose)

Day 30 visit (within 5 days) Draw tacrolimus trough levels, serum creatinine, estimated glomerular filtration rate, serum potassium, and blood glucose. Complete tremor questionnaire with participant.

During or prior to Day 30 visit Oral swab performed to be analyzed for testing of metabolic enzymatic activity (This will be performed to determine ability of the patient to metabolize tacrolimus)

ELIGIBILITY:
Inclusion Criteria:

Adult patient who is 18 years of age or older receiving a kidney transplant at the Temple University Hospital's Kidney Transplant Program who are capable of understanding consent and volunteer to take part in the study

Exclusion Criteria:

Scheduled for multiple organ transplant at enrollment Non-English speaking Pregnant women Moderate-severe hepatic impairment (Child Pugh > 10 or bilirubin > 2) Existing contraindications to tacrolimus-based products including known hypersensitivity to tacrolimus or any other component of the formulation Receiving concomitant medications known to have strong drug-drug interaction potential with tacrolimus including fluconazole, voriconazole, posaconazole, isavuconazole, itraconazole, ketoconazole, diltiazem, verapamil, metronidazole, erythromycin, clarithromycin, rifampin, rifabutin, rifapentine, phenytoin, fosphenytoin, phenobarbital, primidone, carbamazepine, St. John's Wort, efavirenz, neivrapine, etravirine, atazanavir, darunavir, fosamprenavir, indinavir, lopinavir, ritonavir, nelfinavir, saquinavir, tipranavir, cobicistat

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2021-05-23 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Diamond, PharmD, Principal Investigator — Temple University Hospital
Locations (1):
- Temple University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tacrolimus Extended-release 0.13mg/kg/Day
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tacrolimus Extended-release 0.13mg/kg/Day
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 24
  White | 9
  More than one race | 0
  Unknown or Not Reported | 3
History of hypertension [Number; unit: participants] | 28
History of diabetes mellitus [Number; unit: participants] | 9
History of focal segmental glomerulosclerosis [Number; unit: participants] | 1
Calculated panel reactive antibody (%) [Median (Inter-Quartile Range); unit: percentage] | 0 [0 to 10]
Actual body weight (kg) [Mean (Standard Deviation); unit: kg] | 87.4 (18.4)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 30 (5.5)
Deceased donor [Number; unit: participants] | 25
Living Donor [Number; unit: participants] | 11
History of prior transplant [Number; unit: participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to First Therapeutic Tacrolimus Trough Concentration From Initiation of Tacrolimus Extended Release Measured in Days
Description: Therapeutic tacrolimus trough= 8-10ng/mL
Time Frame: Within the first 30 days of kidney transplant
Population: Two participants were not included in the genotype analysis comparison since their genotype samples were unable to be analyzed.
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Non-Expresser: Participant who did not express activity of the CYP3A5 enzyme
- Intermediate Metabolizer: Participant who expressed at least one CYP3A5*1 allele
- Extensive Metabolizer: Participant who expressed two CYP3A5*1 alleles
Arm/Group | Non-Expresser | Intermediate Metabolizer | Extensive Metabolizer
Number analyzed (Participants) | 15 | 13 | 6
days | 4.5 [1 to 7] | 6 [4 to 11.5] | 13.5 [7.5 to 20.25]

2. Secondary Outcome: Average Estimated Glomerular Filtration Rate Within 30 Days
Description: eGFR
Time Frame: 30 days
Population: Kidney transplant recipients
Measure: Median (Inter-Quartile Range); unit: ml/min/173m^2
Arm/Group | Non-Expresser | Intermediate Metabolizer | Extensive Metabolizer
Number analyzed (Participants) | 15 | 13 | 6
ml/min/173m^2 | 40 [27 to 58] | 46 [30 to 58.5] | 31.5 [25 to 56.3]

3. Secondary Outcome: Number of Participants With no Impact of Tremor on Quality of Life
Description: Assessed via QUEST questionnaire which includes a self-assessment of tremor impact on quality of life. The following areas related to impact on tremor are assessed by this scale:
  1. Patients will select the severity of tremor in each of the following body parts on a scale of (none: no tremor at any time, mild: mild tremor not causing difficulty in performing any activities, moderate: tremor causes difficulty in performing some activities, marked: tremor causes difficulty in performing most or all activities, severe: tremor prevents performing some activities).
     * Head
     * Voice
     * Right arm/hand
     * Left arm/hand
     * Right leg/foot
     * Left leg/foot
  2. Several questions will be answered relating to specific situations and the impact of tremor on those situations (scale: never/no, rarely, sometimes, frequently, always/yes, not applicable)
Time Frame: At 30 days after kidney transplant
Population: Kidney transplant recipients
Measure: Count of Participants; unit: Participants
Arm/Group | Tacrolimus Extended-release 0.13mg/kg/Day
Number analyzed (Participants) | 36
Participants | 35

4. Secondary Outcome: Weight-based Tacrolimus Dose During Study Period
Description: Weight-based tacrolimus dose during study period
Time Frame: 30 days
Population: Kidney transplant recipients
Measure: Median (Inter-Quartile Range); unit: mg/kg/day
Arm/Group | Non-Expresser | Intermediate Metabolizer | Extensive Metabolizer
Number analyzed (Participants) | 15 | 13 | 6
mg/kg/day | 0.128 [0.102 to 0.142] | 0.136 [0.108 to 0.169] | 0.176 [0.128 to 0.217]

5. Secondary Outcome: Tacrolimus Dose During Study Period
Description: Tacrolimus dose during study period
Time Frame: 30 days
Population: Kidney transplant recipients
Measure: Median (Inter-Quartile Range); unit: mg/day
Arm/Group | Non-Expresser | Intermediate Metabolizer | Extensive Metabolizer
Number analyzed (Participants) | 15 | 13 | 6
mg/day | 9.6 [9.2 to 10.1] | 12.5 [10.6 to 14.5] | 13.8 [10.4 to 14.4]

6. Secondary Outcome: Tacrolimus Trough Level During Study Period
Description: Tacrolimus trough level during study period
Time Frame: 30 days
Population: Kidney transplant recipients
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Non-Expresser | Intermediate Metabolizer | Extensive Metabolizer
Number analyzed (Participants) | 15 | 13 | 6
ng/mL | 10.78 (2.1) | 9.18 (1.6) | 7.98 (1.3)

7. Secondary Outcome: Weight Based Tacrolimus Dose at Therapeutic Concentration
Description: Weight based tacrolimus dose at therapeutic concentration
Time Frame: At time of therapeutic tacrolimus concentration up to 30 days
Population: Kidney transplant recipients
Measure: Median (Inter-Quartile Range); unit: mg/kg/day
Arm/Group | Non-Expresser | Intermediate Metabolizer | Extensive Metabolizer
Number analyzed (Participants) | 15 | 13 | 6
mg/kg/day | 0.13 [0.12 to 0.165] | 0.20 [0.125 to 0.25] | 0.19 [0.138 to 0.265]

8. Secondary Outcome: Tacrolimus Dose at Therapeutic Tacrolimus Concentration
Description: Tacrolimus dose at therapeutic tacrolimus concentration
Time Frame: At time of therapeutic tacrolimus concentration up to 30 days
Population: Kidney transplant recipients
Measure: Median (Inter-Quartile Range); unit: mg/day
Arm/Group | Non-Expresser | Intermediate Metabolizer | Extensive Metabolizer
Number analyzed (Participants) | 15 | 13 | 6
mg/day | 12 [10 to 14] | 16 [13 to 20] | 16 [11 to 20.5]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Tacrolimus Extended-release 0.13mg/kg/Day
All-Cause Mortality (participants affected / at risk) | 0/36
Serious Adverse Events (participants affected / at risk) | 1/36
Other Adverse Events (participants affected / at risk) | 0/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tacrolimus Extended-release 0.13mg/kg/Day (N=36)
Neurotoxicity (Nervous system disorders) | 1 (1) — Significant tremor

LIMITATIONS AND CAVEATS:
Single-center design Adjustment of LCPT doses in accordance with institution specific guidelines and physician preference Other genotype impact on tacrolimus metabolism not captured in this study (non-CYP3A5 genetic determinants of metabolic activity) Short follow-up period of 30 days Small sample size Open-label design Single-arm design

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/45/NCT03713645/Prot_002.pdf
  • Statistical Analysis Plan (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/45/NCT03713645/SAP_003.pdf